CLINICAL TRIAL: NCT02617589
Title: A Randomized Phase 3 Open Label Study of Nivolumab vs Temozolomide Each in Combination With Radiation Therapy in Newly Diagnosed Adult Subjects With Unmethylated MGMT (Tumor O-6-methylguanine DNA Methyltransferase) Glioblastoma (CheckMate 498: CHECKpoint Pathway and Nivolumab Clinical Trial Evaluation 498)
Brief Title: An Investigational Immuno-therapy Study of Nivolumab Compared to Temozolomide, Each Given With Radiation Therapy, for Newly-diagnosed Patients With Glioblastoma (GBM, a Malignant Brain Cancer)
Acronym: CheckMate 498
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-498; 2015-003739-37 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2015-11-26; First posted 2015-12-01 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Brain Cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — Nivolumab; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Radiotherapy Arm (Experimental): Nivolumab IV infusion + Radiotherapy dose as specified
  Interventions: Drug: Nivolumab; Radiation: Radiotherapy
- Temozolomide + Radiotherapy Arm (Active Comparator): Temozolomide + Radiotherapy dose as specified
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nivolumab
  Arms: Nivolumab + Radiotherapy Arm
Drug: Temozolomide
  Arms: Temozolomide + Radiotherapy Arm
Radiation: Radiotherapy

SUMMARY:
The purpose of this study is to evaluate patients with glioblastoma that is MGMT-unmethylated (the MGMT gene is not altered by a chemical change). Patients will receive Nivolumab every two weeks in addition to radiation therapy, and then every four weeks. They will be compared to patients receiving standard therapy with temozolomide in addition to radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, age ≥ 18 years old
* Newly-diagnosed brain cancer or tumor called glioblastoma or GBM
* Tumor test result shows MGMT unmethylated type
* Karnofsky performance status of ≥ 70 (able to care for self)

Exclusion Criteria:

* Prior treatment for GBM (other than surgical resection)
* Any known tumor outside of the brain
* Recurrent or secondary GBM
* Active known or suspected autoimmune disease
* Biopsy with less than 20% of tumor removed

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (125):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Local Institution - 0083, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Local Institution - 0019, Los Angeles, California
  - Sutter Institute For Medical Research, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - The Regents of the University of California, San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University Of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - The University Of Chicago, Chicago, Illinois
  - University Of Kansas Medical Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Local Institution - 0006, Detroit, Michigan
  - Washington University School OF Medicine-Siteman Cancer Center, St Louis, Missouri
  - JFK Medical Center, Edison, New Jersey
  - Local Institution - 0064, Hackensack, New Jersey
  - Columbia University Medical Center (Cumc), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Preston Robert Tisch Brain Tumor Center at Duke University, Durham, North Carolina
  - Local Institution - 0010, Cleveland, Ohio
  - Local Institution - 0095, Columbus, Ohio
  - Local Institution - 0132, Allentown, Pennsylvania
  - Local Institution - 0007, Philadelphia, Pennsylvania
  - Medical University Of South Carolina, Charleston, South Carolina
  - Local Institution - 0090, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - University Of Texas Md Anderson Cancer Ctr, Houston, Texas
  - Local Institution - 0068, Salt Lake City, Utah
  - Swedish Neuroscience Institute, Seattle, Washington
- Australia (5):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Local Institution - 0003, Heidelberg, Victoria
  - Local Institution - 0004, Prahran, Victoria
  - Local Institution - 0001, Nedlands, Western Australia
  - Local Institution - 0002, New South Wales
- Austria (2):
  - Local Institution - 0061, Linz
  - Local Institution - 0060, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Uz Leuven, Leuven
- Canada (3):
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Denmark (2):
  - Local Institution, Copenhagen
  - Local Institution, Odense
- France (8):
  - Local Institution - 0032, Bron
  - Local Institution, Lille
  - Local Institution - 0024, Marseille
  - Local Institution - 0101, Nancy
  - Local Institution - 0023, Paris
  - Local Institution - 0038, Paris
  - Centre Eugene Marquis, Rennes
  - Local Institution - 0106, Toulouse
- Germany (11):
  - Local Institution - 0051, Bonn
  - Local Institution - 0139, Cologne
  - Local Institution - 0072, Erlangen
  - Local Institution - 0049, Frankfurt am Main
  - Local Institution - 0073, Freiburg im Breisgau
  - Local Institution - 0054, Hamburg
  - Local Institution - 0052, Heidelberg
  - Local Institution - 0138, Munich
  - Local Institution - 0050, Münster
  - Local Institution - 0055, Regensburg
  - Local Institution - 0056, Tübingen
- Israel (2):
  - Local Institution - 0096, Petah Tikva
  - Local Institution - 0097, Tel Aviv
- Italy (6):
  - Local Institution - 0076, Bologna
  - Local Institution - 0079, Milan
  - Local Institution - 0126, Padua
  - Local Institution - 0135, Rozzano (milano)
  - Local Institution - 0078, Siena
  - Local Institution - 0077, Torino
- Japan (21):
  - Local Institution - 0115, Nagoya, Aichi-ken
  - Local Institution - 0125, Chiba, Chiba
  - Local Institution - 0123, Hiroshima, Hiroshima
  - Local Institution - 0122, Sapporo, Hokkaido
  - Local Institution - 0129, Kobe, Hyōgo
  - Local Institution - 0111, Tsukuba, Ibaraki
  - Local Institution - 0121, Kanazawa, Ishikawa-ken
  - Local Institution - 0131, Kagoshima, Kagoshima-ken
  - Local Institution - 0133, Sagamihara-shi, Kanagawa
  - Local Institution - 0119, Kumamoto, Kumamoto
  - Local Institution - 0117, Kyoto, Kyoto
  - Local Institution - 0116, Kyoto, Kyoto
  - Local Institution - 0134, Okayama, Okayama-ken
  - Local Institution, Hirakata-shi, Osaka
  - Local Institution - 0130, Suita-shi, Osaka
  - Local Institution - 0113, Hidaka, Saitama
  - Local Institution - 0128, Bunkyo-ku, Tokyo
  - Local Institution - 0114, Chuo-ku, Tokyo
  - Local Institution - 0118, Mitaka-shi, Tokyo
  - Local Institution - 0110, Yamagata, Yamagata
  - Local Institution - 0112, Tokyo
- Netherlands (4):
  - NKI AVL, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Mc, Rotterdam
  - Local Institution - 0063, Utrecht
- Local Institution, Oslo, Norway
- Poland (2):
  - Local Institution - 0080, Gdansk
  - Local Institution - 0081, Warsaw
- Russia (2):
  - Local Institution - 0070, Moscow
  - Local Institution - 0105, Moscow
- Spain (7):
  - Local Institution, Badalona-Barcelona
  - Local Institution, Barcelona
  - Local Institution - 0028, Barcelona
  - Local Institution - 0029, Madrid
  - Local Institution, Madrid
  - Local Institution, Santiago de Compostela
  - Local Institution - 0025, Valencia
- Sweden (2):
  - Local Institution, Lund
  - Local Institution, Solna
- Switzerland (3):
  - Local Institution - 0059, Geneva
  - Local Institution - 0057, Lausanne
  - Local Institution - 0053, Zurich
- United Kingdom (4):
  - University College Hospital, London, Greater London
  - Christie Hospital Nhs Found. Trust, Manchester, Greater Manchester
  - Royal Marsden Hospital, Sutton, Surrey
  - Beaston West of Scotland Cancer Centre, Glasgow

REFERENCES:
- [Derived] Grkovski M, Daras M, Bale T, Lyashchenko S, Reiner AS, Mellinghoff IK, Schoder H, Dunphy MPS. 18F-BMS-986229 PET imaging of tumor PD-L1 expression in glioblastoma patients. EJNMMI Res. 2025 Sep 26;15(1):124. doi: 10.1186/s13550-025-01283-x. PMID 41003913
- [Derived] Omuro A, Brandes AA, Carpentier AF, Idbaih A, Reardon DA, Cloughesy T, Sumrall A, Baehring J, van den Bent M, Bahr O, Lombardi G, Mulholland P, Tabatabai G, Lassen U, Sepulveda JM, Khasraw M, Vauleon E, Muragaki Y, Di Giacomo AM, Butowski N, Roth P, Qian X, Fu AZ, Liu Y, Potter V, Chalamandaris AG, Tatsuoka K, Lim M, Weller M. Radiotherapy combined with nivolumab or temozolomide for newly diagnosed glioblastoma with unmethylated MGMT promoter: An international randomized phase III trial. Neuro Oncol. 2023 Jan 5;25(1):123-134. doi: 10.1093/neuonc/noac099. PMID 35419607
- [Derived] Woroniecka K, Fecci PE. Immuno-synergy? Neoantigen vaccines and checkpoint blockade in glioblastoma. Neuro Oncol. 2020 Sep 29;22(9):1233-1234. doi: 10.1093/neuonc/noaa170. No abstract available. PMID 32691060
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Radiation Therapy: Nivolumab 240 mg every 2 weeks for 8 doses, then 480 mg every 4 weeks administered intravenously
- Temozolomide + Radiation Therapy: Temozolomide 75 mg/m2 daily during radiation therapy, then 150 mg/m2 Days 1-5 for Cycle 1, then increased to 200 mg/m2 Days 1-5 for Cycles 2-6 administered orally
Period: Randomization
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Started | 280 | 280
Completed | 278 | 275
Not Completed | 2 | 5
Not completed — Request to Discontinue Study Treatment | 1 | 3
Not completed — Participant Withdrew Consent | 1 | 2
Period: Treatment
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Started | 278 | 275
Completed | 0 | 76
Not Completed | 278 | 199
Not completed — Other Reasons | 3 | 3
Not completed — Poor/Non Compliance | 1 | 1
Not completed — Maximum Clinical Benefit | 0 | 2
Not completed — Participant Withdrew Consent | 2 | 6
Not completed — Participant Request to Discontinue | 12 | 21
Not completed — Adverse Event Unrelated to Study Drug | 16 | 9
Not completed — Death | 1 | 1
Not completed — Study Drug Toxicity | 27 | 20
Not completed — Disease Progression | 216 | 136

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized using all randomized subjects (all enrolled subjects who were randomized to any treatment arm)
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy | Total
Number analyzed (Participants) | 280 | 280 | 560
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (10.8) | 56.5 (11.3) | 57.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 105 | 195
  Male | 190 | 175 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 112 | 95 | 207
  Unknown or Not Reported | 165 | 183 | 348
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 231 | 240 | 471
  Black or African American | 4 | 3 | 7
  Asian | 33 | 28 | 61
  Other | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death due to any cause. A participant who has not died will be censored at the last known alive date.
Time Frame: up to 3 years
Population: All Randomized Participants: All enrolled Participants who were randomized to any treatment arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Number analyzed (Participants) | 280 | 280
Months | 13.40 [12.62 to 14.29] | 14.88 [13.27 to 16.13]
Statistical Analysis 1: Comparison: Nivolumab + Radiation Therapy vs Temozolomide + Radiation Therapy; Test type: Superiority — Hazard Ratio is Nivolumab over Temozolomide; p = 0.0037, Log-rank test stratified; Log-rank test stratified by complete or partial resection at baseline as entered into the IVRS; Stratified Cox proportional hazard model = 1.31, 95% CI 2-sided [1.09 to 1.58]

2. Secondary Outcome: Kaplan-Meier Plot of Progression Free Survival
Description: PFS was defined as the time from randomization to the date of the first documented tumor progression or death due to any cause. Participants who did not have disease progression or who did not die were censored at the date of last tumor assessment. Participants who did not have any on study tumor assessment and did not have tumor progression or die were censored at the randomization date. Participants who started any subsequent anti-cancer therapy without a prior reported progression were censored at the last tumor assessment prior to initiation of the subsequent anti-cancer therapy. Participants who had surgical resection post start of study treatment were censored at the last tumor assessment date prior to initiation of surgical resection. PFS was determined by investigator reported response based on the Radiologic Assessment in Neuro-Oncology criteria.
Time Frame: From randomization to the date of the first documented tumor progression or death due to any cause (up to approximately 6 years)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Number analyzed (Participants) | 280 | 280
Months | 6.01 [5.65 to 6.21] | 6.21 [5.98 to 6.90]
Statistical Analysis 1: Comparison: Nivolumab + Radiation Therapy vs Temozolomide + Radiation Therapy; Test type: Superiority — Hazard Ratio is Nivolumab over Temozolomide; Log-rank test stratified; Log-rank test stratified by complete or partial resection at baseline as entered into the IVRS; Stratified Cox proportional hazard model = 1.43, 95% CI 2-sided [1.19 to 1.71]

3. Secondary Outcome: Overall Survival Rate at 24 Months
Description: The overall survival (OS) rate of (nivolumab + radiation therapy) and (temozolomide + radiation therapy) estimated as Kaplan-Meier probability of survival at 24 months. OS was defined as the time between the date of randomization and the date of death due to any cause. A participant who has not died was censored at the last known alive date.
Time Frame: At 24 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Number analyzed (Participants) | 280 | 280
Percentage of participants | 10.6 [7.3 to 14.6] | 21.2 [16.5 to 26.3]

4. Secondary Outcome: Overall Survival in Tumor Mutational Burden (TMB) High Population
Description: OS in all randomized participants that are tumor mutational burden high. OS was defined as the time between the date of randomization and the date of death due to any cause. A participant who has not died was censored at the last known alive date.
Time Frame: From randomization to the date of death due to any cause (up to approximately 6 years)
Population: Data was not and will never be collected
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression Free Survival in Tumor Mutational Burden (TMB) High Population
Description: PFS in all randomized participants that are tumor mutational burden high. PFS was defined as the time from randomization to the date of the first documented tumor progression or death due to any cause. Participants who did not have disease progression or who did not die were censored at the date of last tumor assessment. Participants who did not have any on study tumor assessment and did not have tumor progression or die were censored at the randomization date. Participants who started any subsequent anti-cancer therapy without a prior reported progression were censored at the last tumor assessment prior to initiation of the subsequent anti-cancer therapy. Participants who had surgical resection post start of study treatment were censored at the last tumor assessment date prior to initiation of surgical resection. PFS was determined by investigator reported response based on the Radiologic Assessment in Neuro-Oncology criteria.
Time Frame: as for outcome 2
Population: Data was not and will never be collected
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Number analyzed (Participants) | 0 | 0

6. Post Hoc Outcome: Kaplan-Meier Plot of Overall Survival (OS) - Extended Collection
Description: OS was defined as the time between the date of randomization and the date of death due to any cause. A participant who has not died was censored at the last known alive date. Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date (assessments were made until March 4, 2022).
Time Frame: From randomization to the date of death due to any cause (up to approximately 6 years)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
Number analyzed (Participants) | 280 | 280
Months | 13.34 [12.55 to 14.16] | 14.92 [13.27 to 16.10]
Statistical Analysis 1: Comparison: Nivolumab + Radiation Therapy vs Temozolomide + Radiation Therapy; Test type: Superiority — Hazard Ratio is Nivolumab over Temozolomide; p = 0.0024, Log-rank test stratified; Log-rank test stratified by complete or partial resection at baseline as entered into the IVRS; Stratified Cox proportional hazard model = 1.31, 95% CI 2-sided [1.10 to 1.55]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from the participant's randomization to their study completion (up to approximately 6 years). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy (up to approximately 67 months).
Description: The total number at risk for all-cause mortality represents all participants who were randomized. The total number at risk by any serious adverse event and other (not including serious) adverse events represents all participants that received at least 1 dose of study medication.
Arm/Group | Nivolumab + Radiation Therapy | Temozolomide + Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 269/280 | 253/280
Serious Adverse Events (participants affected / at risk) | 206/278 | 141/275
Other Adverse Events (participants affected / at risk) | 262/278 | 259/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Radiation Therapy (N=278) | Temozolomide + Radiation Therapy (N=275)
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 8
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Visual field defect (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2
Adverse event (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 1
Gait disturbance (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 6 | 3
Impaired healing (General disorders) | 1 | 0
Malaise (General disorders) | 3 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0
Polyserositis (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 2
Sudden death (General disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Encephalitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 2 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 2
Pneumonia aspiration (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 4
Transaminases increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 89 | 57
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 0
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Aphasia (Nervous system disorders) | 4 | 3
Ataxia (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 6 | 8
Cerebellar stroke (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 4 | 1
Epilepsy (Nervous system disorders) | 9 | 11
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 11 | 5
Hemianopia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 9 | 6
Hydrocephalus (Nervous system disorders) | 2 | 1
IIIrd nerve disorder (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 2 | 3
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 2
Neurological decompensation (Nervous system disorders) | 1 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 4 | 1
Seizure (Nervous system disorders) | 37 | 30
Subdural hygroma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Apathy (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 4
Drug dependence (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Testicular disorder (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Euthanasia (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 5
Embolism (Vascular disorders) | 6 | 2
Haematoma (Vascular disorders) | 1 | 2
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Radiation Therapy (N=278) | Temozolomide + Radiation Therapy (N=275)
Anaemia (Blood and lymphatic system disorders) | 16 | 11
Lymphopenia (Blood and lymphatic system disorders) | 7 | 24
Neutropenia (Blood and lymphatic system disorders) | 1 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 26
Hypothyroidism (Endocrine disorders) | 18 | 2
Dry eye (Eye disorders) | 14 | 3
Vision blurred (Eye disorders) | 16 | 4
Abdominal pain (Gastrointestinal disorders) | 16 | 7
Constipation (Gastrointestinal disorders) | 54 | 80
Diarrhoea (Gastrointestinal disorders) | 44 | 23
Nausea (Gastrointestinal disorders) | 66 | 105
Vomiting (Gastrointestinal disorders) | 35 | 63
Asthenia (General disorders) | 25 | 27
Fatigue (General disorders) | 123 | 128
Gait disturbance (General disorders) | 24 | 7
Malaise (General disorders) | 14 | 13
Oedema peripheral (General disorders) | 17 | 15
Pyrexia (General disorders) | 30 | 16
Nasopharyngitis (Infections and infestations) | 21 | 13
Urinary tract infection (Infections and infestations) | 23 | 14
Fall (Injury, poisoning and procedural complications) | 14 | 13
Radiation skin injury (Injury, poisoning and procedural complications) | 30 | 23
Alanine aminotransferase increased (Investigations) | 23 | 20
Lymphocyte count decreased (Investigations) | 15 | 32
Neutrophil count decreased (Investigations) | 3 | 18
Platelet count decreased (Investigations) | 8 | 41
Weight decreased (Investigations) | 20 | 20
White blood cell count decreased (Investigations) | 6 | 15
Decreased appetite (Metabolism and nutrition disorders) | 33 | 50
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 17
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 | 12
Aphasia (Nervous system disorders) | 30 | 20
Cognitive disorder (Nervous system disorders) | 14 | 12
Dizziness (Nervous system disorders) | 41 | 19
Dysgeusia (Nervous system disorders) | 14 | 16
Headache (Nervous system disorders) | 115 | 96
Hemiparesis (Nervous system disorders) | 24 | 12
Memory impairment (Nervous system disorders) | 19 | 14
Seizure (Nervous system disorders) | 35 | 36
Somnolence (Nervous system disorders) | 19 | 8
Anxiety (Psychiatric disorders) | 18 | 9
Confusional state (Psychiatric disorders) | 23 | 14
Depression (Psychiatric disorders) | 22 | 12
Insomnia (Psychiatric disorders) | 29 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 73 | 88
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 22
Rash (Skin and subcutaneous tissue disorders) | 40 | 18
Hypertension (Vascular disorders) | 16 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT02617589/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02617589/SAP_001.pdf